CLINICAL TRIAL: NCT05528757
Title: Limb-Girdle Video Assessment Concept Elicitation and Feasibility Study
Brief Title: Limb-Girdle Video Assessment
Status: Terminated | Type: Observational
Why Stopped: Contract termination/lack of funding
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: Coalition to Cure Calpain 3 (C3) (Unknown); Jain Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CAS-CAS008-01
Record Dates: First submitted 2022-08-24; First posted 2022-09-06 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Limb-Girdle Muscular Dystrophy ; Subtypes 2A, 2B, and 2I
Keywords: Limb-Girdle Muscular Dystrophy; Outcome Measure Development; Video Captures; Remote Assessment; Concept Elicitation; Feasibility Testing
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMDs Patients: Patients with a genetically confirmed diagnosis of a LGMD subtype 2A, 2B, or 2I

SUMMARY:
The purpose of this study is to develop a new remote-based video assessment outcome measure for Limb-Girdle Muscular Dystrophy (LGMD) trials. The overall objectives for this study are: 1. Identify domains and tasks meaningful to participants with a Limb-Girdle Muscular Dystrophy (LGMD) for development of the LGVA, including considerations for subtype heterogeneity and functional subgroup branching; 2. Determine the feasibility and reliability of the LGVA with test-retest of the LGVA Video Capture Manual; 3. Assess and refine the LGVA Video Capture Manual to ensure standardization and incorporate feedback from participants; 4. Collect source material videos using the LGVA Video Capture Manual to support the development of scorecards for the LGVA.

DETAILED DESCRIPTION:
The purpose of this study is to gain insight from people living with an LGMD and gather source material videos to develop and test Limb-Girdle Video Assessment (LGVA), a new outcome measure designed to assess changes in functional abilities of participants in LGMDs clinical trials. The LGVA is being designed as a remote video capture to assess nuanced changes in compensatory movement patterns over time. This study involves two stages. In the concept elicitation stage, the tasks for the LGVA Video Capture Manual will be finalized based on feedback from participants living with an LGMD 2A, 2B, or 2I in various stages of disease progression. After finalizing the LGVA Video Capture Manual, source material videos will be collected to evaluate the feasibility and appropriateness of the LGVA tasks, standardize capture procedures, and inform the development of scorecards for the LGVA.

ELIGIBILITY:
* Person with confirmed diagnosis of an LGMD 2A, 2B, or 2I
* ≥14 years of age at the timing of consent (if age 14 - 17, consent from the parent/ legal guardian is also needed)
* Able to read, speak, and understand English
* Residing in the USA
* Willing and able to complete an electronic survey, which includes questions about personal characteristics and medical history as well as review of tasks
* Willing and able to discuss their experiences as a person living with an LGMD in a group setting
* Willing and able to complete 2 rounds of video capture following instructions in the LGVA Video Capture Manual in a 30-day period
* Willing and able to complete an exit interview to discuss their experiences capturing and recording videos with the LGVA Video Capture Manual

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons living with a confirmed diagnosis of LGMD 2A, 2B, or 2I.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Assessing the fluctuation of movement abilities of LGMDs patients via remote video capture. | January 2023 - March 2023
  Using the newly developed LGVA Video Capture Manual, participants are asked to record two sets of videos of them performing assigned tasks. Participants will have one week to complete each round of video capture, with approximately one month between each round. Videos will be captured remotely and uploaded through a secure platform.

SECONDARY OUTCOMES:
Task Selection Survey | August 2022 - September 2022
  Electronic survey asking LGMDs patients about tasks and activities they perform in their daily life, and if/ how these are impacted by their LGMD symptoms.
Focus Group | September 2022 - October 2022
  Small group discussion of participants with similar functional abilities to discuss the progression of symptoms and heterogeneity among subtypes.
Exit Interview | January 2023 - March 2023
  After the feasibility video captures are complete, participants are asked about their experiences using the LGVA Video Capture Manual and the recording procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Carroll, Study Director — Casimir
Locations (1):
- Casimir, Kingston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No